CLINICAL TRIAL: NCT06693375
Title: A Phase 2a, Exploratory, Two-Part, Open-Label Trial to Evaluate Dose and Safety of NanoEcho Particle-1 (Ferumoxtran) Using NanoEcho Imaging Device Examinations of Rectal Lymph Nodes in Healthy Volunteers, Part A, and Rectal Cancer Patients, Part B.
Brief Title: To Evaluate Dose and Safety of NanoEcho Particle-1 Using NanoEcho Imaging Device Examinations of Rectal Lymph Nodes in Healthy Volunteers and Rectal Cancer Patients.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NanoEcho AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NEIS001; 2024-515335-29-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-12; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteers; Rectal Cancer Patients
MeSH Terms: interventions — Magnetic Iron Oxide Nanoparticles; Contrast Media

STUDY DESIGN:
Intervention Model Description: Part A: In total 12 healthy male participants, or healthy female participants of non-childbearing potential, aged 18 to 50 years (inclusive), with a body mass index (BMI) of 18.5 to 30.0 kg/m2 will be considered for trial participation.
  Part B: Male participants, or female participants of non-childbearing potential, aged >18 years with primary rectal cancer (clinical stage T1-T4) planned for surgery with suspected spread to lymph nodes will be considered for trial participation.
  In Part A, the following dose levels will apply. Each participant will be in one condition. Each condition will be examined by MMUS at 7hours, 24hours, 48hours &72hours post dose:
  * Condition1: Dose 1: 28 mg Fe (7 mg Fe/mL, 4 ml in total )
  * Condition2: Dose 2: 56 mg Fe (3,5 mg Fe/mL, 16 mL in total)
  * Condition3: Dose 2: 56 mg Fe (14 mg Fe/mL, 4 mL in total)
  * Condition4: Dose 3: 112 mg Fe (14 mg Fe/mL, 8 mL in total)
  In Part B, the dose level to be applied will be decided based on the outcome of Part A.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dosing of IMP followed by MMUS evaluation (Experimental): In Part A, Each condition will be evaluated with MMUS after 7hours, 24hours 48hours and 72hours. The following conditions will apply:
  Condition 1: Dose 1: 28 mg Fe (7 mg Fe/mL) Condition 2: Dose 2: 56 mg Fe (3,5 mg Fe/mL) Condition 3: Dose 2: 56 mg Fe (14 mg Fe/mL) Condition 4: Dose 3: 112 mg Fe (14 mg Fe/mL) In Part B, the dose level to be applied as well as the timepoint from MMUS evaluation, will be decided based on the outcome of Part A.
  Interventions: Drug: Iron oxide nanoparticles; Device: Rectal Magnetomotoric ultrasound (MMUS)

INTERVENTIONS:
Drug: Iron oxide nanoparticles — Submucosal injection of nanoparticles in rectum, 28 mg Fe (7 mg Fe/mL)
  Other Names: contrast agent
Device: Rectal Magnetomotoric ultrasound (MMUS) — MMUS examination of lymphnodes in rectum
Drug: Iron oxide nanoparticles — Submucosal injection in rectum 56 mg Fe (3,5 mg Fe/mL)
  Other Names: Contrast agent
Drug: Iron oxide nanoparticles — Submucosal injection in rectum : 56 mg Fe (14 mg Fe/mL)
  Other Names: contrast agent
Drug: Iron oxide nanoparticles — Submucosal injection in rectum 112 mg Fe (14 mg Fe/mL)
  Other Names: contrast agent

SUMMARY:
Clinical nodal staging for rectal cancer tumours in early stages, is today shown to be unreliable and no precise or accurate methods exist. Thus, there is an unmet need for better clinical staging of rectal cancer in early stages. If new imaging techniques for clinical staging of early rectal cancer are developed an opportunity for increased treatment by local excision and decreased unnecessary radical surgery would be possible.

NanoEcho Particle-1 (NEP-1, Ferumoxtran Lyophilisate 20 mg Fe/mL) will be used, in combination with NanoEcho Imaging Device, to enhance the signal in the detection and identification of possible spread of rectal cancer to nearby rectal regional lymph nodes by magnetomotive ultrasound (MMUS) technology.

NEP-1 is an ultrasmall superparamagnetic iron oxide (USPIO)-based contrast agent. It belongs to the specific contrast agents-group, which are specific to reticuloendothelial system (liver, spleen, lymph nodes, bone marrow), mainly represented by iron oxide nanoparticles coated with macromolecules such as dextran in the presence of adjuvants (mineral salts, polyhydric alcohols, etc.). It belongs to the USPIO sub-group (with a mean particle diameter of 30 nm.

The NanoEcho Imaging Device is based on the MMUS technology. It aims to identify possible spread of rectal cancer to nearby rectal regional lymph nodes by visualisation of the movement, generated by the nanoparticles (nTrace).

The iron oxide-based nanoparticles, NEP-1, are administered submucosally at four separate administration sites locally in rectum, close to the suspected tumour area. After some time allowing the particles to spread, the MMUS probe, dressed in a probe cover with ultrasound gel inside, is inserted into the rectum. The nanoparticles are set in motion by a magnetic field, introduced by a rotating magnet located inside the probe. The motion of the tissue, the so-called tissue displacement, is detected with ultrasound and called NanoEcho visualisation of the movement generated by the nanoparticles (nTrace) and is visualised on the screen of the NanoEcho Imaging Device. The higher the concentration of the nanoparticles, the stronger the nTrace signal. Based on the distribution pattern of the particles, the system aims to support the user in distinguishing between healthy and metastatic lymph nodes located nearby the tumour within the rectal region.

Part A In Part A (healthy volunteers) of the trial, NEP-1 will be administered on a single occasion, followed by four MMUS-assessments, in four ascending dose groups of three participants each.

Part B In Part B (rectal cancer patients) of the trial, NEP-1 will be administered on a single occasion, followed by a MMUS assessment in a maximum of ten patients with rectal cancer. The dose level of NanoEcho Particle-1 (Ferumoxtran) to be used and the timepoint for the MMUS assessment will be decided based on Part A.

ELIGIBILITY:
Inclusion Criteria:

Part A

1. Willing and able to give written informed consent for participation in the trial.
2. Healthy male participant, or female participant of non-childbearing potential aged 18 to 50 years, inclusive.
3. Body mass index (BMI) ≥ 18.5 and ≤ 30.0 kg/m2 at the time of the screening visit.
4. Medically healthy participant without abnormal clinically significant medical history, physical findings, vital signs, ECG and laboratory values at the time of the screening visit, as judged by the Investigator. (Discussion is encouraged between the Investigator and the Sponsor Medical Representative regarding the clinical relevance of any abnormal laboratory value during the pre dose period).
5. Women of non-childbearing potential are pre-menopausal females who have undergone any of the following surgical procedures; hysterectomy, bilateral salpingectomy or bilateral oophorectomy, or who are post-menopausal defined as 12 months of amenorrhea (in questionable cases a blood sample with detection of follicle stimulating hormone [FSH] >25 IU/L is confirmatory).

Male participants must be willing to use condom or be vasectomised or practice sexual abstinence from heterosexual intercourse (only allowed when this is the preferred and usual lifestyle of the participant) to prevent pregnancy and drug exposure of a partner and refrain from donating sperm from the administration of IMP until 3 months after the administration of IMP. Any female partner of a non-vasectomised male participant who is of childbearing potential must use contraceptive methods with a failure rate of < 1% to prevent pregnancy (see above) from at least 2 weeks prior to the administration of IMP to 4 weeks after the administration of IMP.

Part B

1. Willing and able to give written informed consent for participation in the trial aged 18 to 99 years, inclusive.
2. Participant with primary rectal cancer planned for surgery with suspected spread to lymph nodes. No suspicion of systemic tumour spread. MRI must have been performed within the last 3 months before administration of IMP.
3. Diagnosed with clinical stage T1-T4.
4. It should be possible to use a probe in rectum (no tumour that blocks).
5. Male participant, or female participant of non-childbearing potential ≥ 18 years of age.
6. Women of non-childbearing potential are pre-menopausal females who have undergone any of the following surgical procedures; hysterectomy, bilateral salpingectomy or bilateral oophorectomy, or who are post-menopausal defined as 12 months of amenorrhea (in questionable cases a blood sample with detection of FSH >25 IU/L is confirmatory).

Male participants must be willing to use condom or be vasectomised or practice sexual abstinence from heterosexual intercourse (only allowed when this is the preferred and usual lifestyle of the participant) to prevent pregnancy and drug exposure of a partner and refrain from donating sperm from the administration of IMP until 3 months after the administration of IMP. Any female partner of a non-vasectomised male participant who is of childbearing potential must use contraceptive methods with a failure rate of < 1% to prevent pregnancy (see above) from at least 2 weeks prior to the administration of IMP to 4 weeks after the administration of IMP.

Exclusion Criteria:

Part A

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the trial, or influence the results or the participant's ability to participate in the trial.
2. Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the administration of IMP.
3. Malignancy within the past 5 years, with the exception of in situ removal of basal cell carcinoma.
4. Any planned major surgery within the duration of the trial.
5. Any previous or current anorectal disorder which may increase risk or burden of trial participation.
6. Any positive result at the screening visit for serum hepatitis B surface antigen, hepatitis C antibodies and/or human immunodeficiency virus (HIV).
7. After 10 minutes supine rest at the screening visit, any vital signs values outside the following ranges: - Systolic blood pressure: <90 or ≥140 mmHg, or - Diastolic blood pressure <50 or ≥90 mmHg, or - Pulse <40 or ≥90 bpm
8. Prolonged QTcF (>450 ms), cardiac arrhythmias or any clinically significant abnormalities in the resting ECG at the screening visit, as judged by the Investigator.
9. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to the IMP, IMP excipients or other parenteral iron products, or excipients of the enema to be used in the trial.
10. Person with pacemaker.
11. Person with metal implants.
12. Previous history of full radiation of rectum.
13. Regular use of any prescribed or non-prescribed medications, including antacids, analgesics, herbal remedies, vitamins and minerals, within 2 weeks prior to the (first) administration of IMP, except occasional intake of paracetamol (maximum 2000 mg/day and not exceeding 3000 mg/week), as well as nasal decongestants without cortisone, antihistamine or anticholinergics for a maximum of 10 days, at the discretion of the Investigator.
14. Planned treatment or treatment with another investigational drug within 3 months prior to Day -1. Participants consented and screened but not dosed in previous phase I trials are not to be excluded.
15. Current smokers or users of nicotine products. Irregular use of nicotine (e.g., smoking, snuffing, chewing tobacco) less than three times/week is allowed before the screening visit.
16. Positive screening result for drugs of abuse or alcohol at the screening visit or on admission to the trial site prior to the (first) administration of the IMP. (Positive results that are expected given the participant's medical history and prescribed medications can be disregarded as judged by the Investigator.)
17. History of alcohol abuse or excessive intake of alcohol, as judged by the Investigator.
18. Presence or history of drug abuse, as judged by the Investigator.
19. History of, or current use of anabolic steroids, as judged by the Investigator.
20. The Investigator considers the participant unlikely to comply with trial procedures, restrictions and requirements.

Part B History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the trial, or influence the results or the participant's ability to participate in the trial.

2. Person with any kind of stoma. 3. Person with pacemaker. 4. Person with metal implants. 5. Previous history of radiation of rectum. 6. Prescence of malignancy other than rectal cancer. 7. After 10 minutes supine rest at the screening visit, any vital signs values outside the following ranges: - Systolic blood pressure: <90 or ≥140 mmHg, or - Diastolic blood pressure <50 or ≥90 mmHg, or - Pulse <40 or ≥90 bpm 8. Prolonged QTcF (>450 ms), cardiac arrhythmias or any clinically significant abnormalities in the resting ECG at the screening visit, as judged by the Investigator.

9. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to the IMP, IMP excipients or other parenteral iron products.

10. Planned treatment or treatment with another investigational drug within 3 months prior to Day -1. Participants consented and screened but not dosed in previous phase I trials are not to be excluded.

11. The Investigator considers the participant unlikely to comply with trial procedures, restrictions and requirements.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Part A: Normalised average nTrace value for all lymph nodes at all timepoints | From dosing and up to 72 hours.
  Dose-response curve and Time-response curve for normalised average nTrace value. nTrace value is NanoEcho visualisation of the movement generated by the nanoparticles
Part B, Normalised average nTrace value for all lymph nodes | From dosing to end of MMUS examination up to 72 hours

SECONDARY OUTCOMES:
Part A. Size of lymph nodes with and without detectable nTrace in Healthy Volunteers | From dosing and up to 72 hours after dosing
  At what size of lymph nodes is (i) lymph nodes detectable (B mode) but no nTrace detectable in lymph nodes? (ii) nTrace detectable in lymph nodes? (iii) nTrace showing an even distribution in lymph nodes?
Part A, Frequency, seriousness, and intensity of adverse events (AEs) for the IMP and the medical device. | From dosing until end of study Day 8 after dosing
Part A. User experience | From dosing up to 72 hours
  Result of user experience questionnaire
Part B. Number of lymph nodes detected by NanoEcho diagnostic method compared to historic MRI data per section and overall | After the MMUS examination up to 72 hours after dosing
Part B, True positive fraction (N+) (sensitivity) and true negative fraction (N0) (specificity) of identified lymph node per section of rectum. | At end of MMUS examination up to 72 hours after dosing
Part A. Distance from injection to lymphnodes with and without detectable nTrace | From dosing and up to 72 hours after dosing
  At what distance from the injection is (i) lymph nodes detectable (B mode) but no nTrace detectable in lymph nodes? (ii) is nTrace detectable in lymph nodes? (iii) is nTrace showing an even distribution in lymph nodes?
Part B. Size of lymph nodes with and without detectable nTrace in Rectal Cancer patients | From dosing and up to 72 hours after dosing
  At what size of lymph nodes is (i) lymph nodes detectable (B mode) but no nTrace detectable in lymph nodes? (ii) is nTrace detectable in lymph nodes? (iii) is nTrace showing an even distribution in lymph nodes?
Part B, Frequency, seriousness, and intensity of adverse events (AEs) for the IMP and the medical device. | From dosing until end of study Day 8 after dosing
Part B. User experience | From dosing up to 72 hours
  Result of user experience questionnaire
Part B. Distance from injection to lymph nodes with and without detectable nTrace in Rectal Cancer Patients | From dosing and up to 72 hours after dosing
  At what distance from the injection is (i) lymph nodes detectable (B mode) but no nTrace detectable in lymph nodes? (ii) is nTrace detectable in lymph nodes? (iii) is nTrace showing an even distribution in lymph nodes?
Part B, Size of detectable metastases | End of MMUS examination up to 72 hours after dosing
Part B, distance form tumour to detectable tumour infiltration | End of MMUS examination up to 72 hours after dosing
Part A, Frequency and nature of device deficiencies (DDs). | From dosing until end of last examination after 72 hours
Part A, Safety and Tolerability of NEP 1 and NanoEcho Imaging Device examination in healthy volunteers. | From dosing until end of study Day 8 after dosing
  Clinically significant changes in vital signs, ECG, safety laboratory measurements (haematology, clinical chemistry, coagulation) and physical examination findings.
Part B, Frequency and nature of device deficiencies (DDs). | From dosing until end of last MMUS examination after 72 hours after dosing
Part B, Safety and Tolerability of NEP 1 and NanoEcho Imaging Device examination in Rectal Cancer Patients | From dosing until end of study Day 8 after dosing
  Clinically significant changes in vital signs, ECG, safety laboratory measurements (haematology, clinical chemistry, coagulation) and physical examination findings.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Consultants, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlies results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact info@nanoecho.se